CLINICAL TRIAL: NCT04745416
Title: Clinical Characteristics of Patients With Hematological Cancer Diagnosed and Severe Acute Respiratory Syndrome Coronavirus 2 Infection at the Hospital de Alta Especialidad de Ixtapaluca and the Hospital General de México "Dr. Eduardo Liceaga"
Brief Title: Clinical Characteristics of Patients With Leukemia and COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Head of the hematology hospitalization area, Hospital General de Mexico
Other Study IDs: DECS/JPO-CT-400-2020
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Leukemia, Acute; Covid19; Leukemia, Lymphoblastic
MeSH Terms: conditions — Leukemia; COVID-19; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leukemia and COVID-19: Patients diagnosed with acute lymphoblastic leukemia according to the criteria of the World Health Organization and confirmed diagnosis of COVID-19 by RT-PCR test
- Leukemia: Patients diagnosed with acute lymphoblastic leukemia according to the criteria of the World Health Organization without suspicion of COVID-19

SUMMARY:
The purpose of this study is to describe the main clinical characteristics of patients with de novo acute lymphoblastic leukemia treated inside the third level hospitals converted to Coronavirus disease 2019 (COVID-19) attention for the metropolitan area of Mexico City.

DETAILED DESCRIPTION:
Retrospective, observational study in patients with diagnosis of acute lymphoblastic leukemia, according to the criteria of the World Health Organization, from April 2020 to December 2020. Patients was cared for in the hematology department of the Hospital Regional de Alta Especialidad de Ixtapaluca or the Hospital General de México. Both hospitals have been assigned as Coronavirus disease 2019 (COVID-19) hospitals, limiting the access, number of outpatient visits and chemotherapy protocols.

Real-time polymerase chain reaction (RT-PCR) test for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was performed for patients with respiratory symptoms or history of contact with suspected / confirmed cases of COVID-19 Upon having a positive RT-PCR test, patients were transferred to a respiratory isolation unit to continue their recovery. Support treatment for COVID-19 was based on local considerations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of acute lymphoblastic leukemia according to the criteria of the World Health Organization.

Exclusion Criteria:

* Age less than 18 years
* Incomplete medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first diagnosis of acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 1 year
Progression free survival | through study completion, an average of 1 year
Number of relapses | through study completion, an average of 1 year
  Cases with more than 5 percent of blasts in bone marrow and as relapse to the central nervous system with the presence of blasts in cerebrospinal fluid
Complete Remission | through study completion, an average of 1 year
  Bone marrow has less than 5 percent blast cells, blood cell counts are within the normal range, and there are no signs or symptoms of leukemia
COVID-19 confirmed | From the date of leukemia diagnosis to the end of the induction chemotherapy cycle 1 (each cycle is 28 days)
  Reactive SARS-CoV-2 RT-PCR test

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Hospital Regional de Alta Especialidad de Ixtapaluca, Ixtapaluca, State of Mexico
  - Hospital General de México "Dr. Eduardo Liceaga", Mexico City